CLINICAL TRIAL: NCT04200794
Title: Formal String Instrument Training in a Class Setting Enhances Cognitive and Sensorimotor Development of Primary School Children
Brief Title: Group Music Practice Enhances Development
Acronym: OC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: James62Ra&D
Record Dates: First submitted 2019-12-05; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Cognitive Change; Motor Activity
Keywords: music-practice; group-setting; randomized-controlled-trial; multiple-transfer-effects; cognitive; sensorimotor; matrix-reasoning; string-instruments
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal cluster RCT (randomized controlled trial) with an intervention group and an active control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- musical instrumental training (Experimental): Bi-weekly musical string instrument training in a group setting, over 24 months, provided by professional string instrument teachers
  Interventions: Behavioral: musical instrumental training
- sensitization to music (Active Comparator): Bi-weekly sensitization to music in a group setting, over 24 months, involving listening, playing small percussive instruments and choir singing, provided by professional school music teachers
  Interventions: Behavioral: sensitization to music

INTERVENTIONS:
Behavioral: musical instrumental training — Learning to play a string instrument in a group setting (school class)
  Other Names: Orchestre en Classe
  Arms: musical instrumental training
Behavioral: sensitization to music — sensitization to music via listening, theory, moderate practice on small percussive instruments and choir singing in a group setting (school class)
  Other Names: Classical school music lessons according to the Swiss school system
  Arms: sensitization to music

SUMMARY:
This randomized controlled trial shows for the first time that focused musical instrumental practice as compared to traditional sensitization to music provokes multiple transfer effects in the cognitive and sensorimotor domain. Over the last two years of primary school (10-12-year-old children), sixty-nine children received biweekly musical instruction in a group setting by professional musicians within the regular school curriculum. The intervention group learned to play string instruments, whereas the control group, peers in parallel classes, was sensitized to music via listening, theory, and some practice. Broad benefits manifested in the intervention group as compared to the control group for working memory, attention, processing speed, cognitive flexibility, matrix reasoning, sensorimotor hand function and bimanual coordination Apparently, learning to play a complex instrument in a dynamic group setting impacts development much stronger than classical sensitization to music. Our results therefore highlight the added value of intensive musical instrumental training in a group setting, encouraging general implementation in public primary schools, better preparing children for secondary school and for daily living activities.

DETAILED DESCRIPTION:
This 2-year longitudinal study compared cognitive and sensorimotor development of two groups of children. Both groups received two music courses of 45 minutes per week in a class setting (maximum 20 children per class), given by professional musicians.

The intervention groups (n=34) learned to play string instruments "Orchestra in Class", the control groups (n=35) followed the standard Swiss school curriculum, with "sensitization to music" lessons, lacking focused instrumental practice.

Children who received protocolled extracurricular music lessons before or during the study, were excluded from the analyses.

The groups were compared at baseline (T0) after one year (T1) and after two years (T2) using standardized psychometric tests, evaluating cognitive and sensorimotor functions as well as tests on musicality.

Music practice, covering a wide and diverse field of skills and abilities, from sensorimotor to cognitive activities at the highest level, is a real driving force for development. Widely distributed regions in the brain, which support all these functions, are trained and better coordinated as a result of this practice. This provokes changes in the morphology and function of the brain. Consequently, practicing music regularly brings benefits that go far beyond musicality. The results of various studies indicate that children who practice music show increased verbal memory, verbal intelligence, reading, visual-spatial processing, executive functions, attention, logical reasoning, and according to some authors even better mathematics or even IQ and social skills.

Available evidence of beneficial musical practice effects on cognitive child development predominantly concerns children of parents with a high socioeconomic and educational background [10] and typically results from private lessons. Additionally, most of the time, the child is interested to learn a musical instrument, inducing a motivational bias. Evaluation of beneficial transfer effects restrains in general to a limited number of capacities or skills and randomized controlled trials (RCTs) with active control groups are scarce.

Here, the investigators compared children who intensively practiced different string instruments in a class setting within a specific Orchestra in Class (OC) program, to peers in parallel classes that received the same amount of musical instruction, also within an entire class, but lacking focused training on a complex musical instrument. Entire existing classes were assigned randomly to the OC and the Control programs (cluster randomization). The study took place in public primary schools in popular neighborhoods in the Geneva area, avoiding confounding music effects with effects of socioeconomic background.

The investigators anticipated that cognitive functions strongly involved in musical practice like working memory, attention, information processing, cognitive flexibility and abstract reasoning, as well as fine sensorimotor function would provoke enhanced positive transfer effects in the OC group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* The experimental group will include students from 2 classes 7P HarmoS (1st year of research) and 8P HarmoS (2nd year of research) who participate in the "Orchestre en classe" program in a public primary school in the vicinity of Geneva.
* The Control group will include students from 2 classes 7P (1st year of research) and 8P (2nd year of research) who do NOT participate in the "Orchestre en classe" program, in the same and a nearby public primary school in the vicinity of Geneva.

HarmoS: primary school education system in French-speaking Switzerland

Exclusion Criteria (both groups)

* hearing deficits;
* development disorders
* epilepsy
* other severe health or neurological problems
* non-consent of the parents or the child
* children who have taken music lessons outside the school curriculum before or during the study will be excluded from the study

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Working memory change | 24 months
  Changed scores at a backward digit span task (WISC-R; Wechsler, 2005).
Executive function change | 24 months
  Changed scores at attention tasks, cognitive flexibility tasks and speed of information processing tasks (D2 Test of Attention; Brickenkamp and Zillmer, 1998);Children's Color Trails Test (CCTT; Llorente, 2003) Higher scores at attention tasks, cognitive flexibility tasks and speed of information tasks processing (D2 Test of Attention; Brickenkamp and Zillmer, 1998); Children's Color Trails Test (CCTT; Llorente, 2003) .
Change in abstract thinking (Matrices subtest of the WISC-IV (Wechsler, 2003)) | 24 months
  Changed scores at a matrix reasoning task

SECONDARY OUTCOMES:
Changed sensorimotor functioning | 24 months
  Changed scores atall 4 subtests of the Purdue Pegboard task (Lafayette, 1999), involving manual dexterity and bimanual coordination

CONTACTS AND LOCATIONS:
Overall Officials: Clara James, PhD, Principal Investigator — School of Health Sciences Geneva
Locations (1):
- School of Health Sciences Geneva; HES-SO University of Applied Sciences and Arts Western Switzerland, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data of this study are deposited on a YARETA, a FAIR digital solution for long-term preservation of research data for all Geneva Universities (https://yareta.unige.ch). DOI: 10.26037/yareta:dhglarpzdfcgzefx4pky7sua3m
Time Frame: As soon as the data are published, I would estimate the embargo at 6 months
Access Criteria: Individual Access will be accredited to known researchers in the field.
URL: https://yareta.unige.ch

REFERENCES:
- Available data/document: Individual Participant Data Set — https://yareta.unige.ch — The data of this study are deposited on a YARETA, a FAIR digital solution for long-term preservation of research data for all Geneva Universities (https://yareta.unige.ch). DOI: 10.26037/yareta:dhglarpzdfcgzefx4pky7sua3m